CLINICAL TRIAL: NCT02666885
Title: Personalised Postoperative Radiochemotherapy in Patients With Head and Neck Cancer and Development of a Multi-parametric Decision Support System for Personalised Medicine in Radiation Oncology
Brief Title: Personalised Postoperative Radiochemotherapy in Patients With Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZPM_Demonstrator_HNC
Record Dates: First submitted 2015-12-10; First posted 2016-01-28 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2018-02

CONDITIONS: Head and Neck Cancer
Keywords: Personalized Medicine; Radiation Oncology; Functional Imaging; Biomarker; Decision Support System; Radiomics
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Integration of PET/MRI in radiotherapy (Experimental): Integration of pretherapeutical PET/MRI in adjuvant radiotherapy
  Interventions: Radiation: Integration of PET/MRI in radiotherapy

INTERVENTIONS:
Radiation: Integration of PET/MRI in radiotherapy — Integration of pretherapeutical PET/MRI in adjuvant radiotherapy

SUMMARY:
The current trial is evaluating the integration of a pretherapeutical FDG-PET/MRI in the adjuvant radiochemotherapy in patients with head and neck cancer. As a secondary hypothesis the intention is to develop of a multi-parametric decision support system for personalised medicine by integrating functional imaging, γH2AX-analysis and genetic information.

ELIGIBILITY:
Inclusion Criteria:

* locally-advanced HNSCC (Oro- and Hypopharynx) stage III and IV without distant metastases
* no contraindications for PET/MRI
* no contraindications for radiochemotherapy
* informed consent
* ECOG PS 0/2

Exclusion Criteria:

* Secondary malignancies that might influence outcome within 2 years after radiochemotherapy of the HNSCC
* previous PET/CT
* induction therapy
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
locoregional progression free survival | 2 years after primary diagnosis
  15% improvement in loco-regional PFS at 2 years through integrtion of pre-operative PET/MR imaging into RT treatment planning

SECONDARY OUTCOMES:
Disease free survival | 2 years after primary diagnosis
Overall survival | 2 years after primary diagnosis
Development of a multi-parametric decision support system | after termination of recruitment and follow up up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Zips, MD, Prof, Principal Investigator — University Hospital Tuebingen, Department of Radiation Oncology, Tuebingen, Germany
Locations (1):
- University Hospital Tübingen, Department of Radiation Oncology, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes